CLINICAL TRIAL: NCT04756336
Title: Proof of Concept Study on LTX-109 as Treatment for Hidradenitis Suppurativa
Brief Title: LTX-109 as Treatment for Hidradenitis Suppurativa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharma Holdings AS (Industry)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20-109-07
Record Dates: First submitted 2021-01-21; First posted 2021-02-16 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Consecutive case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTX-109 treatment (Experimental): Patients are treated with LTX-109 gel, 3% w/w twice daily (morning- evening) by application on active hidradenitis lesions during the intervention period of 6 weeks
  Interventions: Drug: LTX-109 gel, 3% w/w

INTERVENTIONS:
Drug: LTX-109 gel, 3% w/w — The drug is applied to affected lesions according to treatment regimen

SUMMARY:
An Open label Phase II//proof of concept-study to demonstrate if percutaneous application of LTX-109 in a gel vehicle is a safe treatment of Hidradenitis suppurativa and to identify clinical response to intervention, as well to identify if covariates such as age, disease duration, smoking state and BMI influence patient reported measures.

DETAILED DESCRIPTION:
It is unclear whether bacterial colonization in hidradenitis suppurativa/acne inversa (HS) comprises a primary cause, triggering factor or secondary phenomenon of the disease pathogenesis. Studies imply that aberrant immune responses play a role involving both the innate and adaptive immune system, however the clinical picture of HS lesions appears reminiscent of bacterial infection, e.g. due to intense inflammation and malodorous discharge. Recent microbiological studies indicate certain bacterial species are associated with mature HS lesions. It is demonstrated a significant high occurrence of large bacterial biofilms (aggregates > 50 μm in diameter) in tunnels. In total, an array of studies point to a potential involvement of a specific microbiota in the pathogenesis of HS.

The antimicrobial effect of LTX-109 can reduce or eradicate bacterial growth and thus also the inflammatory stimulus of hidradenitis. The antiinflammatory effects of LTX-109 through inhibition of bacterial colonization or infection can prevent rupture and proliferation of follicular material in the dermis. Hidradenitis in more advanced stages can be targeted with this investigational drug. However, it is not reasonable to expect that chronic, longstanding inflammation and sinus formation will heal in six week of intervention. Therefore, patients with most severe activity (Hurley stadium III) or with widespread disease (>5 palm units) will not be included in the study.

The investigator wishes to document whether LTX-109 is an effective compound on hidradenitis. Evidence-based medical treatment of mild disease consists of topical antibiotics (Clindamycin). Systemic antibiotics (Tetracycline) is used for disease that is more widespread. In other parts of Europe, but not recommended in Norway due to the fear of over-usage of Rifampicin, patients who fail to exhibit response to treatment or have a moderate-to-severe disease, systemic Clindamycin 300 in combination with Rifampicin can be given.

Patients failing to exhibit response to treatment options mentioned above or for moderate-to-severe disease, biologic therapy (Adalimumab) can be administered.

Interestingly, Bacterial growth in HS patients has shown a high level of resistance to antibiotics, including rifampicin, clindamycin and tetracyclines, cited as an empiric choice in HS therapeutic guidelines.

Therefore, other treatment options targeting bacteria in HS is warranted.

It would be important to demonstrate whether the lytic peptidomimetic LTX-109 may be effective in the condition as the treatment has apparent benefits, such as a good safety profile, easy self-administered application and no known risk of development of resistance to the Investigational Medicinal Product.

The study will be open label on 16 patients. Treatment will be twice daily application on affected lesions for 6 weeks. Followup after end of treatment will be 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active hidradenitis in the stage I-II according to Hurley's classification.
2. Patients are referred to a dermatology out-patient clinic or patients already in an established treatment program, where there is indication for new or different treatment, or surgical intervention.
3. Patients must have typical affection of the disease of either axillae, groins, and/or perigenital/perianal area
4. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to international guidelines, and national/local regulations.
5. For women in fertile age: Concents to use highly effective contraception until the end of the study

Exclusion Criteria:

1. Patients in need of emergency medical or surgical treatment of hidradenitis
2. Subjects must not have used the following HS treatments within the specified timeframe prior to Baseline Visit:

   1. Systemic therapy for HS, including but not limited to corticosteroids, antibiotics, dapsone or retinoids within 4 weeks
   2. Targeted biologic treatments (refer to within 5 half-lives [if known]) or within 12 weeks, whichever is longer.
   3. Topical treatments with antibiotics, including but not limited to clindamycin within 4 weeks
3. Patients with hidradenitis affecting larger areas (>5 palm units)
4. Patient does not agree to be registered in the national quality register for HS
5. Pregnant or lactating women
6. Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Investigator assessed signs for local reactions to the Investigational Medicinal Product | End point analysis at 6 weeks
  Investigator assessment of signs of local reactions
Patient reported symptoms for local reactions to the Investigational Medicinal Product | End point analysis at 6 weeks
  Patient reported symptoms for local reactions

SECONDARY OUTCOMES:
Change in Investigator assessment of condition from Baseline | End point analysis after 6 weeks
  Investigator assessed change in condition assessed by Hidradenitis suppurativa score (Sartorius) from Baseline to week 6
Change in Investigator assessment disease activity from Baseline | End point analysis after 6 weeks
  Investigator assessed change in disease activity assessed by Hurley's stage division from Baseline to week 6
Change in Investigator assessed number of lesions from Baseline | End point analysis after 6 weeks
  Investigator assessed change in number of inflammatory lesions from Baseline to week 6 assessed by International Hidradenitis Suppurativa Severity Score System
Change in Patient recorded Dermatology Life Quality Index (DLQI) from Baseline | Endpoint analysis at week 6
  Change in patient recorded Dermatology Life Quality Index (DLQI) from Baseline to week 6
Change in Patient recorded Visual Analog Score for pain (VAS) from Baseline | Endpoint analysis at week 6
  Change in patient recorded Visual Analog Score for pain (VAS) from Baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Grimstad, Phd., MD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No